CLINICAL TRIAL: NCT00465179
Title: Phase II Trial of Sunitinib Malate (Sutent) Therapy in Patients With Advanced Non-Clear Cell Renal Cell Carcinoma
Brief Title: Sunitinib Malate in Patients With Non-Clear Cell Renal Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0437; NCI-2010-00583 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-04-20; First posted 2007-04-24 (Estimated); Results first posted 2016-05-04 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-05

CONDITIONS: Renal Cell Cancer; Kidney Cancer
Keywords: Non-Clear Cell Renal Carcinoma; Non-clear cell renal cell cancer; Renal Cell Cancer; Kidney Cancer; Papillary; Chromophobe; Collecting duct carcinoma; CDC; Renal medullary carcinoma; RMC; Sunitinib Malate; Sutent; SU011248
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sunitinib Malate (Experimental): Sunitinib Malate 50 mg by mouth daily for 4 weeks, then 2 weeks off.
  Interventions: Drug: Sunitinib Malate

INTERVENTIONS:
Drug: Sunitinib Malate — 50 mg by mouth daily for 4 weeks, then 2 weeks off.
  Other Names: Sutent; SU011248

SUMMARY:
The goal of this clinical research study is to learn the effectiveness of Sutent® (sunitinib malate, SU011248) in the treatment of patients with non-clear cell renal cell cancer. The safety of sunitinib malate will also be studied.

DETAILED DESCRIPTION:
Sunitinib malate is designed to block pathways that control important events such as the growth of blood vessels that are essential for the growth of cancer.

If you are found to be eligible to take part in this study, you will take sunitinib malate once a day (either with or without food) for 4 weeks in a row followed by 2 weeks of rest with no study drug. These 6 weeks are considered 1 cycle of study treatment.

Around Day 15 of each cycle, your vital signs will be measured and recorded, and you will have blood drawn (about 2 teaspoons) for routine testing. These evaluations can be done at your local doctor's office.

You will be required to return to clinic for a follow-up visit around Day 29 of Cycle 1.

At this visit, your medical history will be recorded, and your ability to perform daily activities will be evaluated. You will have a physical exam, including measurement of your vital signs. You will be asked about any side effects you may have experienced since your last visit. You will be asked about any medicines you may be currently taking. You will have blood drawn (about 4 teaspoons) for routine testing.

Beginning Day 1 of Cycle 3, you will return to clinic every 12 weeks (Day 1 of each cycle). You will have the same evaluations as you did at the Day 29 visit.

On Day 1 of every other cycle, you will have an ECG and a doppler echocardiogram or multigated acquisition (MUGA) scan to evaluate your heart health.

You will have follow-up imaging scans (CT and/or MRI) to track your response to treatment on Day 1 of the first 2 cycles and every 12 weeks thereafter for as long as you are receiving treatment on this study.

You will continue to receive treatment on this study, unless your disease gets worse, you develop an illness that prevents you from continuing treatment, or you experience any intolerable side effects of the study drug. You will be removed from this study if any of these circumstances occur.

This is an investigational study. Sunitinib malate has been authorized by the FDA for treatment of clear cell renal carcinoma. Its use in non-clear cell renal carcinoma is experimental. Up to 60 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed advanced non-clear cell of one of the following subtypes: papillary, chromophobe, collecting duct carcinoma (CDC), renal medullary carcinoma (RMC), or unclassified. Patients with conventional-type renal cell carcinoma who have >/= 20% sarcomatoid component in their primary tumor are eligible. Patients who have sarcomatoid features in fine-needle aspiration (FNA) or core biopsy of any metastatic site are eligible.
2. Patients must have measurable disease.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
4. Patients must have adequate organ and marrow function within 14 days prior to study entry as defined: Hemoglobin >/= 9 g/dl, absolute neutrophil count >/= 1,500/microliter (microL), platelets >/= 100,000/microL, total bilirubin </= 1.5 mg/dl, AST(SGOT) and/or ALT (SGPT) </= 2.5 X institutional uln, except in known hepatic metastasis, wherein may be </= 5 x uln, serum creatinine </= 4 X uln (as long as patient does not require dialysis).
5. Patients must have recovered from any effects of surgery.
6. Female patients of childbearing potential (not postmenopausal for at least 12 months and not surgically sterile) must have a normal plasma beta human chorionic gonadotropin (betaHCG) within 24 hours prior to enrolling in the study.
7. Patients of child fathering or childbearing potential must agree to practice a form of medically acceptable birth control while on study (barrier method, hormonal methods, etc.).
8. Patients must give written informed consent prior to initiation of therapy, in keeping with the policies of the institution. Patients with a history of major psychiatric illness must be judged (by the treating physician) able to fully understand the investigational nature of the study and the risks associated with the therapy.
9. Patients with brain metastases may participate in this trial.
10. Patients who have had up to two prior systemic therapies are eligible to participate in this trial but they should not have had prior Multi-Tyrosine Kinase Inhibitors such as sorafenib or sunitinib malate.

Exclusion Criteria:

1. No prior malignancy is allowed, except for non-melanoma skin cancer, in situ carcinoma of any site, or other cancers for which the patient has been adequately treated and disease free for 2 years.
2. Pregnant or lactating women are excluded.
3. Patients must not be scheduled to receive any experimental drug for MRCC while on study. Patients are permitted to be on concomitant bisphosphonates. Patients are permitted to receive hematopoietic growth factors according to American Society of Clinical Oncology (ASCO) guidelines.
4. Patients must not have had prior radiotherapy to areas of measurable disease, unless they have clearly progressive disease in this site, or there is measurable disease outside the area of prior radiation. Radiotherapy, if needed for palliation, must have been completed at least 2 weeks prior to enrollment on this study.
5. Patients may not have any significant medical disease (other than the malignancy) that, in the investigator's opinion, would increase the risk for participation. Examples of exclusion: unstable angina pectoris, New York Heart Association (NYHA) Grade II or greater congestive heart failure, unstable symptomatic cardiac arrhythmias requiring medication (subjects with controlled chronic atrial fibrillation are eligible), myocardial infarction within 6 months, uncontrolled HTN (blood pressure >150/90 on therapy), corrected QT interval (QTc) interval > 500msec or other significant ECG abnormalities or uncontrolled DM.
6. Patients must not have history of other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of sunitinib malate or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications.
7. Concomitant treatment with drugs with dysrhythmic potential (terfenadine, quinidine, procainamide, disopyramide, sotalol, probucol, bepridil, haloperidol, risperidone, and indapamide) is not recommended.
8. Patients unwilling to participate or unable to comply with the protocol for the duration of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2007-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nizar M. Tannir, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were enrolled between March 2007 and August 2010 at The University of Texas (UT) MD Anderson Cancer Center (MDACC).
Pre-assignment Details: 61 participants were enrolled to the study. 4 participants did not receive any treatment, resulting in 57 participants available for evaluation.
Groups:
- Sunitinib Malate: Sunitinib Malate 50 mg by mouth daily for 4 weeks, then 2 weeks off. These 6 weeks are considered 1 cycle of study treatment.
Period: Overall Study
Arm/Group | Sunitinib Malate
Started | 57
Completed | 4
Not Completed | 53
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 2
Not completed — Progression of Disease | 47

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 57
Age, Continuous [Median (Full Range); unit: years] | 57 [22 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 38
Region of Enrollment [Number; unit: participants]
  United States | 57

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response to Treatment
Description: Response was assessed using Response Evaluation Criteria In Solid Tumors (RECIST). Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least 30% decrease in sum of the longest dimensions (LD) of all target lesions, taking as reference the baseline sum of LD. Stable Disease (SD): Insufficient shrinkage to qualify for partial response, or insufficient increase to qualify for progressive disease, taking as reference the smallest sum longest diameter since the treatment started. Progressive Disease (PD): At least a 20% increase in the sum of LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Every 6 weeks for the first two cycles, then every 12 weeks, up to 2 years
Population: Two participants were not evaluable as one was taken off study due to adverse event and the other due to withdrawal of consent.
Measure: Number; unit: participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 55
participants
  Complete Response | 0
  Partial Response | 3
  Stable Disease | 29
  Progressive Disease | 23

2. Primary Outcome: Median Progression-Free Survival (PFS)
Description: Median Progression-Free Survival was calculated as the time from the date of the first treatment to the date of disease progression or date of death, or the last date of the outcome evaluation, whichever came first.
Time Frame: Every 6 weeks for the first two cycles, then every 12 weeks, up to 2 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 55
months | 2.7 [1.4 to 5.4]

3. Secondary Outcome: Median Overall Survival
Description: Overall survival was estimated using the Kaplan-Meier method.
Time Frame: Baseline till participant death or end of follow-up period, assessed every 6 weeks for the first two cycles, then every 12 weeks, up to 5 years.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 57
months | 16.8 [10.7 to 26.3]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) and Serious Adverse Events (SAEs) were collected from administration of study drug on day 1 of course 1 and on day 1 of all subsequent courses, up to 5 years.
Description: Overall collection period: March 2007 to February 2015.
Arm/Group | Sunitinib Malate
Serious Adverse Events (participants affected / at risk) | 57/57
Other Adverse Events (participants affected / at risk) | 57/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib Malate (N=57)
Fatigue (General disorders) | 16 (16)
Hypertension (Cardiac disorders) | 16 (16)
Neutropenia (Blood and lymphatic system disorders) | 11 (11)
Pain (General disorders) | 7 (7)
Mucositis/Stomatitis (Gastrointestinal disorders) | 6 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5)
Anemia (Blood and lymphatic system disorders) | 5 (5)
Leukopenia (Blood and lymphatic system disorders) | 3 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Sensory Neuropathy (Nervous system disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3)
Anorexia (Gastrointestinal disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Motor Neuropathy (Nervous system disorders) | 1 (1)
Hemorrhage (Vascular disorders) | 1 (1)
Nonneutropenic Fever (General disorders) | 1 (1)
Left Ventricular Diastolic Dysfunction (Cardiac disorders) | 1 (1)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Transaminitis (Hepatobiliary disorders) | 1 (1)
Elevated Lipase (Metabolism and nutrition disorders) | 1 (1)
Myocardial Infarct (Cardiac disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Thrombosis/Embolism (Blood and lymphatic system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Hand-Foot Skin Reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 39 (39)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Sickle-Thalassemia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib Malate (N=57)
Activated Partial Thromboplastin Time Prolonged (Blood and lymphatic system disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 19 (44)
Alkaline Phosphatase (Metabolism and nutrition disorders) | 20 (33)
Allergic Rhinitis (Immune system disorders) | 2 (3) — Including sneezing, nasal stuffines, and postnasal drip
Allergy/Immunology-Other (Immune system disorders) | 1 (1)
Alanine Aminotransferase (Metabolism and nutrition disorders) | 17 (21)
Amylase (Metabolism and nutrition disorders) | 7 (11)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Anorexia (Gastrointestinal disorders) | 17 (23)
Aspartate Transaminase (Metabolism and nutrition disorders) | 31 (50)
Autoimmune Reaction (Immune system disorders) | 3 (6)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 11 (18)
Bruising (Skin and subcutaneous tissue disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 4 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 11 (28)
Cardiac General-Other (Cardiac disorders) | 1 (1)
Cardiac Troponin I (Cardiac disorders) | 1 (1)
Hypercholesteremia (Metabolism and nutrition disorders) | 13 (20)
Confusion (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 24 (34)
Constitutional Symptoms (General disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (18)
Creatine Phosphokinase (Metabolism and nutrition disorders) | 1 (1)
Creatinine (Metabolism and nutrition disorders) | 35 (104)
Creatinine Increased (Metabolism and nutrition disorders) | 2 (8)
Cystitis (Renal and urinary disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 5 (6)
Depression (Nervous system disorders) | 1 (1)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 9 (10)
Diarrhea (Gastrointestinal disorders) | 33 (170)
Dizziness (Nervous system disorders) | 3 (3)
Xerostomia (Gastrointestinal disorders) | 1 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 3 (4)
Dysesthesia (Nervous system disorders) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 3 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 30 (65)
Edema: Head and Neck (Blood and lymphatic system disorders) | 5 (8)
Edema: Limb (Blood and lymphatic system disorders) | 19 (37)
Edema (Blood and lymphatic system disorders) | 2 (3)
Edema: Trunk/Genital (Blood and lymphatic system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Erectile Dysfunction (Reproductive system and breast disorders) | 1 (1)
Fatigue (General disorders) | 52 (311)
Fever (General disorders) | 1 (1)
Fever (General disorders) | 2 (2) — In the absence of neutropenia
Flatulence (Gastrointestinal disorders) | 1 (1)
Gamma-Glutamyl Transpeptidase (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 23 (68)
Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 11 (16)
Headache (Nervous system disorders) | 10 (15)
Heartburn (Gastrointestinal disorders) | 15 (29)
Hemoglobin (Metabolism and nutrition disorders) | 52 (212)
Hemolysis (Blood and lymphatic system disorders) | 3 (3)
Hemorrhage, GI (Vascular disorders) | 1 (1)
Hemorrhage, GU (Vascular disorders) | 3 (5)
Hemorrhage, Pulmonary/Upper Respiratory (Vascular disorders) | 1 (1)
Hemorrhage/Bleeding-Other (Vascular disorders) | 7 (15)
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 6 (9)
Hypertension (Cardiac disorders) | 35 (78)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 16 (23)
Hyperuricemia (Metabolism and nutrition disorders) | 12 (16)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 9 (19)
Hyponatremia (Metabolism and nutrition disorders) | 8 (27)
Hypotension (Cardiac disorders) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 2 (2)
Infection (Infections and infestations) | 8 (9) — With normal ANC or Grade 1 or 2 neutrophils
Infection (Infections and infestations) | 3 (3) — With Grade 3 or 4 neutrophils
Infection-Other (Infections and infestations) | 5 (5)
Insomnia (General disorders) | 2 (4)
Left Ventricular Diastolic Dysfunction (Cardiac disorders) | 3 (4)
Leukocytes (Blood and lymphatic system disorders) | 40 (172)
Lipase (Metabolism and nutrition disorders) | 9 (12)
Lymphatics-Other (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 4 (6)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Memory Impairment (Nervous system disorders) | 2 (2)
Mood Alteration (Nervous system disorders) | 7 (7)
Mucositis/Stomatitis (Gastrointestinal disorders) | 41 (139)
Musculoskeletal and Connective Tissue Disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (2)
Nail Changes (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 41 (149)
Neuroendocrine: ACTH Deficiency (Endocrine disorders) | 1 (1)
Neuropathy: Motor (Nervous system disorders) | 7 (11)
Neuropathy: Sensory (Nervous system disorders) | 19 (54)
Neutrophils/Granulocytes (Blood and lymphatic system disorders) | 24 (119)
Non-Cardiac Chest Pain (General disorders) | 1 (1)
Pain in Extremity (General disorders) | 3 (8)
Pain-Other (General disorders) | 38 (157)
Abdominal Pain (General disorders) | 11 (23)
Back Pain (Musculoskeletal and connective tissue disorders) | 13 (21)
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Chest Pain (General disorders) | 3 (4)
Face Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Oral Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Scalp Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Throat Pain (General disorders) | 1 (1)
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Hypoparathyroidism (Endocrine disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 9 (13)
Platelets (Blood and lymphatic system disorders) | 31 (63)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 5 (15)
Proteinuria (Metabolism and nutrition disorders) | 16 (26)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4)
Pulmonary Hypertension (Cardiac disorders) | 1 (2)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 2 (3)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 28 (44)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) — Dermatitis associated with radiation
Rash: Hand-Foot Skin Reaction (Skin and subcutaneous tissue disorders) | 22 (59)
Renal Failure (Renal and urinary disorders) | 1 (1)
Serum Glutamic Oxaloacetic Transaminase (Metabolism and nutrition disorders) | 1 (1)
Serum Glutamic Pyruvic Transaminase (Metabolism and nutrition disorders) | 1 (1)
Small/Large intestine (Gastrointestinal disorders) | 2 (4)
Syncope (Nervous system disorders) | 1 (1)
Sweating (General disorders) | 2 (2)
Surgical and Medical Procedures (Surgical and medical procedures) | 1 (1)
Taste Alteration (Gastrointestinal disorders) | 18 (26)
Thromboembolic Event (Blood and lymphatic system disorders) | 1 (2)
Thrombosis (Vascular disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 5 (5)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blurred Vision (Eye disorders) | 5 (5)
Flashing Lights/Floaters (Eye disorders) | 1 (1)
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Vomiting (Gastrointestinal disorders) | 28 (85)
Watery Eye (Eye disorders) | 16 (32)
Weight Loss (General disorders) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes